CLINICAL TRIAL: NCT06107985
Title: To Develop and Validate a Structured Exercise Protocol and to Assess Its Effectiveness in Patients With Sub Acromial Impingement Syndrome
Brief Title: To Develop and Validate a Structured Exercise Protocol and Its Efficacy in Sub Acromial Impingement Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Seth Gordhandas Sunderdas Medical College (Other)
Responsible Party: Principal Investigator, Reshma Shashank Gurav, Physiotherapy Specialist, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRC-01-22-428; EC-OA-94-2022 (Other: Seth G.S. Medical College and KEM Hospital, Mumbai,India)
Record Dates: First submitted 2023-10-01; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Subacromial Impingement; exercise protocol; SPADI
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured exercise group (Experimental): Group A (Experimental Group) will receive structured exercises protocol, will be given approximately for two days per week for twelve weeks.
  Interventions: Other: Structured exercise program
- Conventional Exercise group (Active Comparator): Group B (control group) will receive conventional exercise program for two days per week for twelve weeks.
  Interventions: Other: Conventional Exercise Program

INTERVENTIONS:
Other: Structured exercise program — This intervention will be based on shoulder kinetic control, load modification exercises and lumbopelvic stabilization with core stability exercises which is not a part of conventional exercise program for shoulder impingement syndrome patients.
  Arms: Structured exercise group
Other: Conventional Exercise Program — Conventional exercise program for shoulder impingement syndrome patients
  Arms: Conventional Exercise group

SUMMARY:
Shoulder impingement syndrome (SIS) is responsible for 44% to 60% of medical consultations related to shoulder pain with an approximate prevalence of 70-200 per 1000 adults, which implies a remarkable use of health care resources. The cost for society is high and patients with shoulder disorders account for 20% of all disability due to musculoskeletal disorder. The underlying mechanisms are thought to include inflammation, degeneration of the tendons or bursa, dysfunctional scapulothoracic and glenohumeral mechanics, debilitated scapular musculature, joint capsule irregularities, postural abnormalities of the neck and shoulder, and morphological abnormalities of the relevant skeletal elements. There is a need for well-designed structured exercise program in detail considering content, dosage and progression to guide treatment for patients with sub acromial pain.

The purpose of this study is to develop and validate a structured exercise protocol and to assess its effectiveness in patients with sub-acromial impingement syndrome. Through the extensive literature review, the exercise program would be proposed. In Phase 1, We will develop and validate a structured exercise programs for sub acromial impingement syndrome using an expert consensus Delphi-based survey technique. In phase 2, a randomized controlled trial will be conducted. Group A (Experimental Group) will receive newly structured exercises for twelve weeks and Group B (control group) will receive conventional exercise program for 12 weeks. Evaluation of the participant will be done at the baseline using Constant Murley Score, shoulder pain and disability Index (SPADI). Shoulder range of motion, shoulder muscles extensibility will be assessed and scapulothoracic ratio will be calculated and documented. T-FAST test will be conducted to score the patients functional performance.

Assessment will be done at baseline, 3, 6, 9, and 12 weeks in both the groups. At the end of the study the data will be collected, coded and tabulated using descriptive and inferential statistics.

DETAILED DESCRIPTION:
Shoulder pain is very common with an annual population prevalence of up to 46.7%, and a lifetime prevalence of up to 67%.1 In primary care, shoulder pain is the third most common musculoskeletal presentation. 1, 2 Shoulder pain may have an unfavourable outcome, with only about 50% of all new episodes of shoulder complaints presenting in physiotherapy practice showing a complete recovery within 6 months. Symptoms may be disabling in terms of the patient's ability to carry out daily activities at home and at the workplace. The most frequent shoulder diagnosis is subacromial pain syndrome, affecting about half of all shoulder patients, both in general practice and in secondary care. Shoulder impingement syndrome (SIS) is responsible for 44% to 60% of medical consultations related to shoulder pain implies a remarkable use of health care resources. The cost for society is high and patients with shoulder disorders account for 20% of all disability due to musculoskeletal disorder. The diagnosis of SIS is therefore mainly based on functional aspects and on an affected anatomical structure and requires a thorough history and clinical examination, including aspects such as activity and participation restrictions, aggravating and easing factors, or the "patients' perspective on the situation". Physiotherapy assessment has a very significant role to find out the structural and functional impairments and accordingly set the goals of management. Diagnosing the cause and identifying the source or affected structure is of utmost importance in Physiotherapy management. Apart from focusing only on structures, physiotherapy assessment emphasizes on movement dysfunctions and biomechanical derangements commonly seen in patients with impingement. Correction of the biomechanical faults would off load the sub acromial space and reduce the pain. The technique used to correct the biomechanics is called "load modification or Shoulder symptom modification process" and involves techniques: Alterations to thoracic kyphosis, Scapular positioning techniques, Humeral head positioning procedures and pain and symptom neuromodulation procedure. Current evidence for the physiotherapeutic treatment of SIS, summarized in systematic reviews through the last years, supports the specific and structured exercise program. Furthermore, these studies used either different types of exercises in their groups as a basic treatment, or applied a pre-defined set of manual techniques to all patients without considering the individual situation of the patient. Reasons for the selection or the combination of the exercises or the manual techniques used varied considerably between studies, were often not explained and thus remained unclear. Recent systematic review and meta-analysis conducted by Louis Pieter and Jeremy Lewis in 2020 concluded that continued research is needed to more fully understand the uncertainty around the optimal type, dose, and duration of exercise for sub-acromial shoulder pain. Thus, nearly all current systematic reviews emphasize the need for more high quality trials of physiotherapy interventions to optimize the dosimetry of exercise program. The term conventional physiotherapy is uninterpretable and inconclusive especially because there is presumption of how exactly the exercise program is formed. Many of the exercise program do not provide adequate information of what and why interventions are used. There are many varieties of exercises with different rationale and techniques. Hence, it is mandatory to have an adequate description of techniques making up the intervention and rationale for dosage is essential i.e. the number of sessions, intensity, and duration of intervention as per the TIDieR checklist (Template for Intervention description and replication). There is a need for well-designed structured exercise program in detail considering content, dosage and progression to guide treatment for patients with sub acromial pain. This demands developing a specific guidance on how exercise interventions should be reported in clinical trials depending on what structure is affected in intrinsic and extrinsic mechanisms of subacromial impingement syndrome. 4 The purpose of this study is to develop and validate a structured exercise protocol and to assess its effectiveness in patients with sub-acromial impingement syndrome. Through the extensive literature review, the exercise program would be proposed. We will develop and evaluate a structured exercise programs for sub acromial impingement syndrome using an expert consensus Delphi-based survey technique. Structured exercise program will be formed as per the guidelines of TIDieR items which will include the name of the intervention; intervention rationale for essential elements; intervention materials and details about how to access them; description of the intervention procedures; details of intervention providers; mode of delivery of intervention; location of intervention delivery and key infrastructure; details about the number, duration, intensity, and dose of intervention sessions; details of any intervention tailoring; any intervention modifications throughout the study; and details of intervention assessment, monitoring, and level achieved. This intervention will be based on shoulder kinetic control, load modification exercises and lumbopelvic stabilization with core stability exercises which is not a part of conventional exercise program for shoulder impingement syndrome patients. The study will be conducted in two phases. Phase 1 will be to develop and validate a structured exercise program and phase 2 is to evaluate efficacy of structured exercises on pain, range of motion and shoulder functions using Constant Murley score and Shoulder Pain and Disability Index (SPADI) and functional performance using timed functional arm and shoulder test. A randomized controlled trial will be conducted. Group A (Experimental Group) will receive structured exercises for twelve weeks and Group B (control group) will receive conventional exercise program for 12 weeks. Evaluation of the participant will be done at the baseline using Constant Murley Score, shoulder pain and disability Index (SPADI). Shoulder range of motion, shoulder muscles extensibility will be assessed and scapulothoracic ratio will be calculated and documented. T-FAST test will be conducted to score the patients functional performance. Assessment will be done at baseline, 3, 6, 9, and 12 weeks in both the groups. At the end of the study the data will be collected, coded and tabulated using descriptive and inferential statistics. The data will be analyzed to see the efficacy of newly developed structured exercise program versus conventional exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18-60 years
* Symptoms for more than three weeks
* Main complaints in the gleno humeral joint region or the proximal arm
* Presence of one of the following signs indicating SAIS: Neer impingement test, Hawkins-Kennedy impingement test, painful arc with active abduction or flexion. Pain with one of the following resistance tests: external rotation, internal rotation, abduction

Exclusion Criteria:

* Severe pain; pain is > 7/10 on NRS (0 = no pain)
* Shoulder surgery on affected shoulder
* Traumatic shoulder dislocation/ fracture within the past 3 months
* Previous rehabilitation for this episode of shoulder pain
* Reproduction of shoulder pain with active or passive cervical motion
* Systemic inflammatory joint disease
* Global loss of passive shoulder ROM, indicative of adhesive capsulitis
* Full-thickness rotator cuff tear
* Incompetent adults
* Subjects unable to consent
* Patients who are unfit to undergo the suggested exercises as per the protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Score | Baseline, 3, 6, 9, and 12 weeks
  This score is a shoulder-specific assessment tool containing objective measures (range of movement and shoulder strength) and subjective measures (activity of daily living and pain). This scale assesses four aspects related to shoulder pathology; two subjective: pain and activities of daily living (ADL) and two objectives: range of motion (ROM) and strength. The subjective components can receive up to 35 points and the objective 65, resulting in a possible maximum total score of 100 points (best function). Pain and ADL are answered by the patient; ROM and strength require a physical evaluation and are answered by the physiotherapist.
Visual analouge Scale | Baseline, 3, 6, 9, and 12 weeks
  The visual analogue scale (VAS; 0-10) is used to assess the patient's perceived pain intensity at rest, during arm activity and at night during the previous 24 hours at each follow-up. The visual analogue scale (VAS) uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end. Patients are asked to mark a point on the line that best represents their pain. The distance from 'no pain' to the patient's mark is then measured and this equals the Visual Analouge scale score.
The Shoulder Pain and Disability Index (SPADI) | Baseline, 3, 6, 9, and 12 weeks
  The Shoulder Pain and Disability Index is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. To answer the questions, patients place a mark on a 10cm visual analogue scale for each question. Verbal anchors for the pain dimension are 'no pain at all' and 'worst pain imaginable', and those for the functional activities are 'no difficulty' and 'so difficult it required help'. The scores from both dimensions are averaged to derive a total score. The means of the two subscales are averaged to produce a total score ranging from 0 (best) to 100 (worst).
Timed Functional Arm and Shoulder Test | Baseline, 3, 6, 9, and 12 weeks
  The Timed Functional Arm and Shoulder Test (TFAST)is a simple battery of physical performance tests for functional task used for shoulder assessment.

SECONDARY OUTCOMES:
Scapulothoracic ratio Measurement | Baseline, 3, 6, 9, and 12 weeks
  Scapulothoracic ratio is measured with inclinometer to quantify scapular upward rotation associated with varying amounts of humeral elevation for measurement of scapular upward rotation

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Gurav, Principal Investigator — Hamad Medical Corporation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ludewig PM, Cook TM. Alterations in shoulder kinematics and associated muscle activity in people with symptoms of shoulder impingement. Phys Ther. 2000 Mar;80(3):276-91. PMID 10696154
- [Result] Shire AR, Staehr TAB, Overby JB, Bastholm Dahl M, Sandell Jacobsen J, Hoyrup Christiansen D. Specific or general exercise strategy for subacromial impingement syndrome-does it matter? A systematic literature review and meta analysis. BMC Musculoskelet Disord. 2017 Apr 17;18(1):158. doi: 10.1186/s12891-017-1518-0. PMID 28416022
- [Result] Kromer TO, de Bie RA, Bastiaenen CH. Effectiveness of individualized physiotherapy on pain and functioning compared to a standard exercise protocol in patients presenting with clinical signs of subacromial impingement syndrome. A randomized controlled trial. BMC Musculoskelet Disord. 2010 Jun 9;11:114. doi: 10.1186/1471-2474-11-114. PMID 20534140
- [Result] Pieters L, Lewis J, Kuppens K, Jochems J, Bruijstens T, Joossens L, Struyf F. An Update of Systematic Reviews Examining the Effectiveness of Conservative Physical Therapy Interventions for Subacromial Shoulder Pain. J Orthop Sports Phys Ther. 2020 Mar;50(3):131-141. doi: 10.2519/jospt.2020.8498. Epub 2019 Nov 15. PMID 31726927
- [Result] Worsley P, Warner M, Mottram S, Gadola S, Veeger HE, Hermens H, Morrissey D, Little P, Cooper C, Carr A, Stokes M. Motor control retraining exercises for shoulder impingement: effects on function, muscle activation, and biomechanics in young adults. J Shoulder Elbow Surg. 2013 Apr;22(4):e11-9. doi: 10.1016/j.jse.2012.06.010. Epub 2012 Sep 1. PMID 22947240

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT06107985/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT06107985/ICF_001.pdf